CLINICAL TRIAL: NCT00155506
Title: Molecular Genetic Study of Schizophrenia: Parent-Offspring Trios
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 14553; NHRI-CN-MA-9006S
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2002-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Niacin; Genotyping; candidate gene; one proband, normal parents and one normal sibling
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Schizophrenia is a chronic and devastating major psychiatric disorder. Family, twin, and adoption studies indicated that schizophrenia has a significant genetic component. The mode of transmission is still not clear and a multilocus model was proposed. The location of susceptibility gene of schizophrenia is still under active search using molecular genetic methods.

We propose to collect genomic DNA and lymphoblast cell lines of a total of 150 DSM-IV schizophrenic patients and their first degree relatives including parents (parent-offspring trios) and non-affected siblings in three years. Adequate statistical power of molecular genetic studies is a great concern. For this concern, we will examine the patients and their parents clinically by using the Diagnostic Interview for Genetic Studies (DIGS) for diagnostic assessment, and by using neuropsychological battery including sustain attention, executive function, verbal memory and general intelligence for neuropsychological evaluations.

The project is feasible because (1) The PI and his research team have experience in successfully collecting co-affected sib-pair families of schizophrenia and in setting-up molecular genetic laboratory in the past decade. We are experienced and competent to execute this project. (2) The PI and his research team have established the instruments using to clarify the phenotypes including the DIGS, the neuropsychological battery these years.

Major goals of this project are: (1) to cooperate with this important Taiwan Genotype Consortium proposed by the NHRI; (2) to detect major schizophrenia susceptibility genes related to the neuropsychological endophenotype; (3) to do further fine mapping on suggestive linkage markers to replicate previous linkage studies results using our previously-collected co-affected sib-pair family sample; and (4) to deposit the lymphoblast cell lines into NHRI Cell Bank serving as a national resource for basic research in Taiwan.

DETAILED DESCRIPTION:
1. Specific Aims We propose to collect genomic DNA and lymphoblast cell lines of a total of 150 families with the probands fulfilling the criteria of DSM-IV schizophrenia in three years. The first degree relatives of the probands, including parents (parent-offspring trios) and non-affected siblings, a total of about 3 to 6 subjects, will also be recruited in study. Adequate statistical power of molecular genetic studies is the great concern. For this concern, we will examine the probands and family members clinically by using the Diagnostic Interview for Genetic Studies (DIGS) for diagnostic assessment, and using neuropsychological battery including sustain attention, executive function, verbal memory and general intelligence.

   This specific aims of this project are: (1) to cooperate with this important Taiwan Genotyping Consortium proposed by the NHRI; (2) to detect major schizophrenia susceptibility genes which are related to the neuropsychological endophenotype; (3) to do further fine mapping on suggestive linkage chromosome regions to replicate previous linkage studies results using our previously-collected co-affected sib-pair family sample; and (4) to deposit the lymphoblast cell lines into NHRI Cell Bank serving as a national resource for basic research in Taiwan.
2. Background

   1. Genetic Basis of Schizophrenia Most family studies confirm that schizophrenia and related disorders is a familial disorder and that the risk to first degree relatives of schizophrenic patients is approximately ten times the risk to relatives of controls. Twin studies have found concordance rates from 46%~53% for MZ twin pairs, and from 14%~15% for DZ twin pairs (Kendler KS 1983; Gottesman II 1993; Prescott and Gottesman II, 1993); thus provide strong evidence for an hereditary component to schizophrenia. However, the concordance rates in MZ twins is far from 100% , which also emphasizes the importance of environmental factors in the etiology of schizophrenia. The evidence of genetic contribution to the etiology of schizophrenia is further supported by adoption study. Adoption studies of schizophrenia have shown that when biological offspring of schizophrenic mothers were raised by adoptive parents, they showed higher rates of schizophrenia as adults, compared to control adoptees.

   Segregation analyses indicate that multifactorial polygenic model, which posit a large, unspecified number of loci to combine additively in causing schizophrenia, better fit the observed patterns of schizophrenia in family studies than do single major locus model. It was suggested that several genes of small effect in epistasis might responsible for genetic etiology of schizophrenia.

   The location of susceptibility gene of schizophrenia is still under active search using molecular genetic methods. This way of approach included linkage analysis, candidate genes association study, and positional candidate gene approach, there is no a priori hypothesis that would lead one to focus on any given chromosomal region. Thus, the whole genome needs to be systemically screened. A few genome-wide scans of schizophrenia have been published for the decade and many chromosome regions showed suggestive evidences for linkage, including chromosome 1q21-q22, 1q31-q42, 2p22-q21, 4q24-q32, 6p24-p22, 6q16-q23, 8p24-p21, 10p14-p13, 13q14-q32, 15q13-q14, 22q11-q13. However, only a few chromosome regions were ever reported to have genome-wide significant linkage evidences, including chromosome 1q21-q22, 6p24-p22, 8p21 and 13q32.

   Candidate genes studies revealed inconsistent results in the past decade. Neurotransmitter related genes, such as dopamine (D1, D2, D3, D4, D5), serotonin, r-aminobutyric acid and Glutamate receptor genes had been studied using both association and linkage studies and no consistent results obtained. Neuron growth related genes, phospholipase genes, and a potassium channel gene (hKCa3/KCNN3) have been reported association with schizophrenia. The hypothesis about the pathophysiological mechanism of schizophrenia provide the probable candidate genes approach in the molecular genetic study. There exists two issues to be resolved for candidate gene approach using case-control design. Firstly, a critical issue in assessing the significance of association with phenotypic measures is the likelihood of type I errors. Since many genes and phenotypes can be evaluated for schizophrenia, the significance level needs to be adjusted due to the low prior probability and multiple testing. Secondly, the effects of different population admixture between cases and controls may inflate the type I errors Positional candidate gene approach using linkage dysequilibrium strategy may resolve the above two problems raised by the approach of candidate gene association study basing upon the previous linkage results to increase the prior probability and using parent-offspring trios as internal control. This approach is more powerful than linkage study to locate the susceptibility genes of complex disorder as schizophrenia. With the fine mapping linkage evidences, the whole genome sequence and single nucleotide polymorphism (SNP) map, and the advancing microarray technique available, this approach is more efficient to locate the susceptibility genes of schizophrenia. Recently, a study using above strategy has been reported significant linkage dysequilibrium evidence of schizophrenia to a microsatellite polymorphism and a SNP of a gene, NOTCH4 gene, at chromosome 6p21.

   Considering the potentials of positional candidate gene approach using linkage dysequilibrium strategies, we propose to collect parent-offspring trios of schizophrenia as the sample of further molecular genetic study of schizophrenia. With our previous and ongoing efforts in linkage studies of schizophrenia using co-affected sib-pairs of schizophrenia (see preliminary results), this sample can be used for further positional candidate gene studies.

   3. Neuropsychological Deficit in Schizophrenia In the domain of neuropsychology, schizophrenia have been shown to have unique pattern of impairments in central executive function, sustained attention and working memory were rather unique in schizophrenia and are suggestive of frontostriatal dysfunction. It was agreed by most researchers that neuropsychological impairments of schizophrenia were best demonstrated by comprehensive test batteries tapping on various neuropsychological process, rather than single, isolated test and at present, the impairments strongly suggested dysfunction of frontal-temporal-limbic circuit.

   Among the neuropsychological deficits in schizophrenia, visual sustained attention measured by the Continuous Performance Test (CPT) and executive function measured by the Wisconsin Card Sorting Test (WCST) were studied more thoroughly. Common features of the CPT are that participants must respond to predesignated targets among stimuli that are presented at a rapid fixed rate. The discrimination vigilance task of the CPT may consist of a single stimulus (CPT-X, single character or number as the target ) or two successive stimuli (CPT-AX, a character or number preceded by another character or number as the target). The difficulty level of the CPT can be raised further by blurring the stimuli (degraded CPT) or using a relative target (CPT-Identical Pairs Version or CPT-IP). The different CPT versions might tap on different components of sustained attention: the more difficult ones are stable vulnerability indicators, while the simpler ones might be mediating vulnerability indicators in schizophrenia. Among studies specifically examining the relationships between CPT performance indexes and clinical symptom dimensions, one of the most consistent findings is that CPT deficits are associated with negative symptoms. Many studies also found that poorer performance on the CPT were associated with thought disorder or disorganized symptoms.

   Executive function deficits measured by WCST referred to abnormal function of prefrontal cortex. Deficits in WCST performance are enduring and core features of schizophrenia, and predict long term disability, independent of other cognitive deficits. Functional neuroimaging studies have found that the WCST activates the dorsolateral prefrontal cortex and that the dopamimetic drugs improves performance on this task in patients with schizophrenia and enhance the signal to noise of the prefrontal physiological response.

   Previous studies confirmed that deficits in sustained attention and executive function are specific to schizophrenia and related to schizophrenic pathophysiological process. The deficits have also been associated with genetic risk of schizophrenia and may serve as an endophenotype in genetic analysis in schizophrenia.

   4. Endophenotype Approach in Molecular Genetic Studies of Schizophrenia To resolve the problems of insufficient power of genetic analyses and genetic heterogeneity of schizophrenia, an alternative strategy was advocated that the use of a specific neurobiological characteristic of the illness as an additional phenotype that might reflect more closely the effect of a single genetic alteration.

   The visual sustained attention deficits as measured by CPT was an potential endophenotype of the genetic susceptibility to schizophrenia. CPT deficits were present not only in schizophrenia patients, but also in their non-psychotic relatives. Using data from 148 non-psychotic relatives and 345 community adults found that the recurrence risk ratio λwas greater than 15 for the undegraded CPT and greater than 30 for the degraded CPT.

   The executive function deficits as measured by WCST may also serve as an endophenotype in genetic studies of schizophrenia. WCST deficits presented both in schizophrenic patients and their healthy siblings.

   Thus, using CPT deficits and WCST deficits as endophenotypes of schizophrenia would provide a valuable measure of genetic risk, would improve the power of genetic analyses and may help identify susceptibility genes for schizophrenia.

   This endophenotype strategy has been successful in mapping of a neurophysiological deficit of schizophrenia, decrease of P50 inhibition, to loci at chromosome 15q13-14, recently. The genome-wide linkage analysis of the P50 inhibition deficit in nine multiplex schizophrenia families found a significant lod score (Z = 5.30,  = 0) at a loci chromosome 15q14. When the clinical diagnosis of schizophrenia was used as the affected phenotype, the maximum lod score at the same marker was not statistically significant. The other neurobiological deficit, eye tracking dysfunction of schizophrenia has been mapped to chromosome 6p23-21 with the maximum multipoint lod score of 4.02. Again, while the clinical diagnosis of schizophrenia was used as the affected phenotype, the linkage result was non-significant.

   In summary, with our preliminary studies in linkage analyses using co-affected sib-pairs of schizophrenia and neuropsychological deficits in schizophrenia, this project to collect schizophrenics of parent-offspring trios with well-defined neuropsychological endophenotypes, is considered to be one crucial project for searching the susceptibility genes of schizophrenia.
3. Preliminary Studies

   1. Collection of Schizophrenia Co-affected Sibpairs Family The P.I. has been committed himself in collecting the schizophrenia co-affected sib-pairs family since 1990. With the awareness of the importance and critical necessity of diagnostic assessment, these probands, co-affected sib and available non-affected sib as well as the parents were assessed with a semi-structured psychiatrist diagnostic interview using diagnostic criteria of DSM-III-R and/or DSM-IV. Besides, under the evolutionary theoretical model of psychopathology, developmental data were also collected. All these clinical data and family-tree data were established in the data bank of the molecular genetic laboratory (DBMGL) in the Department of Psychiatry, College of Medicine, National Taiwan University under the auspice of the P.I. In total, there are around 120 schizophrenia co-affected sib-pairs families available for linkage analysis in the DBMGL. As a rule, the DNA samples were obtained from the peripheral white cells of all available subjects of the family, especially the co-affected sibs, at least one non-affected sib and the parents. In total, around 1000 DNA samples were in the DBMGL. Cell-lines of EBV-958 transformed lymphoblast cells were established too. All these study subjects were well informed for this study and informed consent obtained. All families participated in this study were invited to join a "New-Hope Family Club" for periodic meeting and discussion. Around 150 schizophrenia cases who received detail clinical assessment and regular follow-up and comprehensive neuropsychological assessment, including CPT, WCST, WAIS-R, and WMS, were recruited for obtaining DNA samples. Around 200 normal control subjects were also recruited for obtaining DNA samples.

      The instruments used in genetic studies have been established. The Diagnostic Interview Schedule for Genetic Study (DIGS) and schizotypy interview schedule (SIS) were translated and modified to be useful in Taiwan subjects. The Perceptual aberration scale (PAS) and Schizotypal personality questionnaire (SPQ) were also used in community study on schizophrenia-related personality disorders. The cross-cultural consideration was employed.

      A 5-year nation-wide collaborative work in Taiwan (Taiwan Schizophrenia Linkage Study, TSLS), sponsored by the NIMH, U.S.A., to collect families with co-affected sib-pairs with schizophrenia has been going on in the third years. A total of 600 families will be collected. DNA samples, cell-lines and clinical data of DIGS, FIGS, as well as neuropsychological testing data were collected. The DNA sample would be open to research teams all over the world.
   2. Molecular Genetic Studies of Schizophrenia Our molecular genetic studies of schizophrenia were supported by three consecutive projects: the molecular genetic project sponsored by the National Science Council (1989-1992), the molecular genetic project of MPGRP (1993-1998) and the molecular genetic project of MPSS (1998-2001) sponsored by NHRI. The early phase (1989-1992) of this molecular genetic project focused on establishing laboratory facilities and collecting co-affected schizophrenic sib-pair families. The 2nd phase of this molecular genetic project (1993-1998) continued the collection of families, and the collection was extended to collect the co-affected bipolar sib-pairs, schizophrenic cases and normal controls. We found the polymorphism of androgen receptor gene of (CAG)n had a probable association with schizophrenia. This finding supported the finding of DeLisi et al. The molecular genetic methods of linkage analysis and candidate gene association were promoted, this laboratory of the P.I. (Dr. Hwu) moved to emphasize in this area too. The results of this laboratory were: (1) The polymorphism of (48bp) repeats in DRD4 receptor gene was not significantly linked with schizophrenia; (2) A single mutation in DRD2 was found not to be associated with schizophrenia (3) The samples of the data bank of this project had joined three international collaboration studies using positional cloning approach which need relatively large sample. The one is organized by Gill et al entitled as "Schizophrenia Collaborative Linkage Group", another was led by Dr. Moises in Kiel University, Germany and the third one is with Dr. Powell in London. All these results revealed the possible markers in chromosomes 6p, 11q, 13q, 19q and 22q. This suggests that Taiwanese patients may have possible susceptibility genes in these regions, except chromosome 13q, fitting an oligogenetic model. (4) The association study on 5-HT2 receptor gene located on chromosome 13q was found to be negative; (5) Clinical epidemiological analysis using co-affected sib-pairs demonstrated the tendency of 3 independent symptom clusters of reality disorganization, disorganization and negative state. (6) Weak linkage evidence to loci at chromosome 6p24-22.

      The 3rd phase of the molecular genetic study (1998-2001) continued focusing at collecting co-affected schizophrenic sib-pair families and linkage analysis on reported suggestive evidences of chromosome regions, including chromosome 1q21-q22, 1q31-q42, 8p24-p21, 15q13-q14, 22q11-q14. The linkage results were (1) suggestive evidence of linkage for schizophrenia with and without the negative symptoms on chromosome 6p24 and 22q12 (2) no linkage evidence of GABAA receptor α1 (GABRA1) , β1 (GABRB1) andβ3 (GABAB3) subunit gene with schizophrenia (3) no linkage evidence of Glutamate GluR5 and GluR6 receptor gene with schizophrenia (4) no linkage evidence of SCA1 gene with schizophrenia (5) suggestive linkage evidence on markers of chromosome 8p with schizophrenia (Hwu et al., 2001a) (6) weak linkage evidence of markers of chromosome 1q31-42 with schizophrenia (7) suggestive linkage evidence of markers on 15q13-14 with schizophrenia (8) modest linkage evidence of schizophrenia to loci at chromosome 1q21-22. The candidate gene approach has revealed the following results: (1) possible association between Dopamine D4 receptor (DRD4) gene polymorphism with quick treatment response of schizophrenia (Liu et al., 2001d) . (2) no association between cytosolic phospholipase A2 (c-PLA2) gene polymorphism and schizophrenia.
   3. Studies on Neuropsychological Deficits in Schizophrenia We found impaired sustained attention by continuous performance test (CPT) as the trait marker of schizophrenia. Family studies have indicated that sustained attention deficits as measured by the CPT are vulnerability markers of schizophrenia. The results are: (1) a substantial proportion of non-psychotic relatives of schizophrenia probands (19-34%) have CPT deficits, which can be predicted from their probands' CPT performance; (2) subjects with schizotypal personality features also exhibit CPT deficits, which are specifically associated with negative factors of schizotypy; (3) CPT deficits are present in schizophrenic patients, are particularly associated with negative and disorganized symptoms, and those with more difficult CPT versions are not amenable to neuroleptic treatment.

   The specificity of CPT was studied in a group of schizophrenia patients (n=41) in contrast to the group of bipolar patients with psychotic symptoms (n=46) and the group of bipolar patients without psychotic symptoms (n=22) and a group of patients with non-psychotic major depressive disorder (n=22). It was found that CPT deficits are stable vulnerable indicators of schizophrenia, mediating vulnerability indicators for bipolar disorder, and state-dependent indicator for major depression. These results demonstrate that CPT deficits are valid trait marker of schizophrenia.

   All these preliminary data support that the PI and his associates is capable in executing this project including collection of parent-offspring trios families, DNA extraction and cell culture laboratory techniques, and the neuropsychological assessment.
4. Research Design and Methods

   1. Subjects We prepare to collect parent-offspring trios families from the Medical Center of National Taiwan University Hospital and the affiliated psychiatric hospitals, the Taoyuan Psychiatric Center. The proband cases to be recruited are the residents of the Northern part of Taiwan. Informed consent will be obtained before the recruitment for study. The first degree relatives to be recruited are the parents and at least one of the unaffected siblings. The diagnosis of the proband cases is of schizophrenia defined by DSM-IV criteria.
   1. Clinical Assessment Measures I. The Diagnostic Interview for Genetic Studies (DIGS) All subjects will be personally interviewed with the DIGS, which was created by Tsuang and Faraone from the NIMH Human Genetics Initiative. The DIGS makes a detailed assessment of the course of illness, and makes a careful assessment of substance abuse and mood symptoms. This allows for an easier differential diagnosis between schizophrenia and substance related psychoses, schizoaffective disorders and psychotic mood disorders. This detailed assessment helps protect against false positive diagnosis.

      In addition, the DIGS provides a rich description of many domains of psychopathology: somatization, major depression, mania/hypomania, dysthymia/depressive personality/hyperthymic personality, alcohol abuse disorders, pathological gambling, and antisocial personality disorder. It also collects self-reported demographic and medical history data. Ratings are also made on the Global Assessment Scale and the Scales for the Assessment of Positive and Negative Symptoms. Schizotypal and other Axis II Cluster A personality features are assessed by using a modified version of the Structured Interview for Schizotypy.

      II. The Family Interview for Genetic Studies (FIGS) As an additional source of pedigree information, the FIGS will be conducted with all members of the family. This interview systematically questions an informant about the presence of psychiatric illness in relatives. We administer the FIGS in three steps. First, the structure of the family pedigree is drawn and reviewed with the informant. Next, psychiatric screening questions are asked about all relatives in the pedigree. Then based on the responses to the screening questions, one or more of five symptom checklists (depression, mania, substance abuse, psychosis, paranoid /schizoid/ schizotypal personality disorder) are completed for each first-degree relative, spouse, or other relative well known to the informant.

      The DIGS and FIGS were translated into Chinese. The reliability and validity have been established in our preliminary studies.

      III. The Diagnostic Procedure All diagnoses will be made using DSM-IV. These diagnoses will be made by two board certified psychiatrists with clinical and research experience in the diagnosis of psychotic patients. Final diagnoses of probands and relatives will be based on the content of the interview, the case vignette, information provided by relatives and a complete review of the medical record by each diagnostician. If the two diagnosticians disagree about any of the patient's diagnoses, a third diagnostician will be used as a tie-breaker.

      IV. Training of Interviewers The training program will certify the interviewers: (1) establish a working knowledge of the diagnostic systems used in the DIGS and FIGS; (2) develop expertise in the administration and scoring of the structured diagnostic instrument; and (3) fully understand the process of informed consent and the need for strict adherence to consent procedures.

      The training program is divided into two stages: (1) formal didactic training and (2) supervised experience using the structured diagnostic interview.

      The didactic training begins with trainees reading and familiarizing themselves with the diagnostic systems used by the DIGS. This initial exposure is supplemented by lectures which review diagnostic criteria for all psychiatric disorders covered by the interview. Central issues addressed in these lectures are: (1) the importance of establishing diagnoses on the basis of objective behavioral description; (2) careful delineation and differentiation of syndromes which involve both psychotic and affective phenomena; and (3) clarification of major differences in syndrome definition among diagnostic systems.

      The second component of training focuses on the structured diagnostic instruments. Trainees first gain familiarity with the structure of the interview. This is facilitated by having trainees conduct practice interviews in which they alternately play the roles of interviewer and subject. These initial interviews are conducted with a senior psychiatrist in attendance to identify problem areas in administration and to ensure clinically sensitive use of the interview.

      The training program also includes a module on the modified Structured Interview for Schizotypy (SIS). The SIS training includes a review of the literature about schizotypal personality disorder, an orientation and review of the instrument, an opportunity for trainees to observe and make clinical ratings of a live interview, and a review and discussion of clinical ratings to clarify scoring criteria. All the training courses have been well established in our preliminary studies.
   2. Neuropsychological Evaluations

      Considering the complexity of the proposed neuropsychological deficits in schizophrenia, a test battery tapping multiple aspects of cerebral process is chosen to explore patients' overall pattern of neuropsychological deficits. The battery consists of tests supposed to measure:
      1. Sustained attention (the Continuous Performance Test (CPT), both in undegraded and degraded test situations)
      2. Central executive functions (Wisconsin Card Sorting Test (WCST); Trail-making B);
      3. Memory function (Weschler Memory Scale-third edition, WMS-III).
      4. Test for general intellectual achievements (block design; picture completion; information; similarity; arithmetic; digit span; digit symbol substitution).

      The neuropsychological test used in present study and validity of the test battery have been well established in our preliminary studies. We prepare to administer the neuropsychological test battery to the probands and all the recruited family members as possible. The neuropsychological test battery is rather time-consuming, estimated to take 3 to 4 hours to complete. Hence, the neuropsychological test battery will be administrated in divided sessions, completed in two days. Two master degree research assistants majored in psychology will perform all the tests.

   2. Laboratory Work: This project has two lines of laboratory work
   1. Collection of blood samples and extraction of DNA Twenty to thirty ml of venous blood will be obtained from all study subjects into purple top and green top vacutainer tubes. The blood sample in purple top tubes will be used for DNA extraction. We prepare to extract the DNA using a modified salting-out method.
   2. Cell-line set-up All blood samples newly collected will have the lymphocyte transformed into lymphoblastic cell for preservation of cell-line which will be deposited into the cell bank of NHRI as the proposal requested. The detail procedures of cell culture established in our molecular genetic laboratory are listed as attached files molecular genetic study.

   3. Data Management We have already set up the computerized DIGS database software in our previous study (Taiwan Schizophrenia Linkage Study, TSLS) and neuropsychological databank in another previous study (Multidimensional Psychopathological Study for Schizophrenia, MPSS). All the clinical and neuropsychological data in this project will be incorporated into these databanks.

   The family pedigree data, DNA data, and cell culture data will be incorporated into our previously established databank: Bank of Molecular Genetic Laboratory Data (BMGLD). This BMGLD will include 4 sets of Data: (1) family tree and genotyping data bank. These data are set-up using the cyrillic program ; (2) DNA sample bank; (3) clinical data and endophenotype bank and (4) cell-line bank. This well organized BMGLD will be of great value for continous research work.

   The data entry procedures will follow the guidelines that we use for our ongoing projects. These procedures seek to maximize the accuracy of data. The data will be double-entered, and the original and verification files will be compared for discrepancies. All datasets will be backed up to disc regularly. The backup and original data sets will be maintained in different locked offices.

   The datasets in this project will be available to other investigators following the guidelines of the RFA. We will create a dataset which will include all data required by the RFA and whatever additional data the NHRI desires to incorporated into the Cell Bank. These data will be sent to the data management center designated by the NHRI for subsequent distribution to the member of genotyping consortium.
5. Anticipated Results We anticipate through this project to attain the following goals: (1) to cooperate with this important Taiwan Genotyping Consortium proposed by the NHRI, (2) to detect major schizophrenia susceptibility genes which are related to the neuropsychological endophenotype, (3) to do further fine mapping on suggestive linkage chromosome regions to replicate previous linkage studies results using our previously-collected co-affected sib-pair family sample, and (4) to deposit the lymphoblast cell lines into NHRI Cell Bank serving as a national resource for basic research in Taiwan.
6. Human Subjects This is a genetic study, all subjects recruited will present his signed informed consent before being enrolled for study. There is no invasive procedure of potential hazard in the process of the clinical interview and the neuropsychological evaluations. Blood samples of 30 c.c. will be drawn. This will be done using a needle and this may cause some painful sensation which is usually negligible in clinical setting. These participating subjects will be reassured as any discomfort feeling happens during the study procedures.

   All researchers participated in this study procedure are all well trained. If these is any unexpected emotional or physical reaction happens during the study procedure, the P.I. of the project should be informed and necessary actions will be taken immediately. Since this is a genetic study, in the study procedure, there may have the genetic counseling issue raised. The participating researchers will be educated before attending this study for this topic of genetic counseling. These subjects or their family who are in need of specific genetic counseling will be refer to the special clinic, locating in the outpatient department of the National Taiwan University Hospital, of the P.I. of this project for special care.
7. Animal Investigation not involved.
8. Potential Hazards The clinical interview, the neuropsychological evaluations, and the blood sample drawn will be very safe. However, this genetic study might provoke some emotional reaction of the family, especially regarding the genetic heritability. In this case, the attending researchers, well trained, will give immediate assurance and assessment. If anything considered to be necessary, these subjects will be referred to the special clinic of the P.I. of this project for special psychiatric care.

The procedure of blood sample drawing might create mild degree of painful sensation or fearful feeling. These cases will be reassured immediately. Generally speaking, this study procedure is safe and the potential hazards is minimal and is manageable if anything happen.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV schizophrenic patients and their first degree relatives including parents (parent-offspring trios) and non-affected siblings

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-11; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University